CLINICAL TRIAL: NCT01118494
Title: Study of Urinary Angiotensinogen as a Marker to Warn the Deterioration of Renal Function in CKD Patients Early.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: HuaShan Hospital of Fudan University, Nephrology Department
Other Study IDs: 08dz1900603
Record Dates: First submitted 2010-04-26; First posted 2010-05-06 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-04

CONDITIONS: Chronic Kidney Disease; Urinary Angiotensinogen
Keywords: CKD; RAS; AGT
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum plasma urine supernatant urine sediment
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CKD patients: People who have been diagnosed with CKD，and been in the stage of 3 or 4.

SUMMARY:
Chronic kidney disease (CKD) that results in end-stage renal disease (ESRD) is a major international health problem. Many clinical markers such as urine protein or eGFR(evaluated glomerular filtration rate),can estimate the renal function, but not sensitive. As well-known, the crucial role of angiotensin II (AngII), the major effector of the renin-angiotensin system (RAS), in the development of renal fibrosis that results in ESRD is widely recognized.Abundant researches find that intrarenal RAS takes an important role on the progression of CKD. At present, no clinical marker is available to evaluate intrarenal AngII activity because it is difficult to measure it directly in patients. So find and establish a bio-marker of local renal RAS activation maybe a breakthrough in early detection and treatment of CKD. Angiotensinogen(AGT) is the only known substrate for renin and the level of AGT in humans is close to Km value for renin. Thus , changes in AGT levels can control the activity of the RAS, and its up-regulation may lead to activity of Ang levels. Then we hypothesis that the AGT is a early bio-marker of local renal RAS activation as well as CKD.

DETAILED DESCRIPTION:
1. Screening: Select CKD(3-4) patients from outpatients, Urine routine examination and Renal B-mode ultrasonography and so on.
2. Confirm: Sign consent with the patients who meet the inclusion criteria, then these patients are included in the study.
3. Create patients records and complete related-inspections.
4. Clinical follow-up: Follow-up once every six months, and we will record every patient's disease progress every time. Each follow-up, the patient needs to leave 5 ml blood samples and 20 ml of urine samples, used for the following study.
5. Detection, Observation and Evaluation: Patients are divided into two groups according to AGT levels: higher than the normal group and the normal group. Observe the changes in eGFR of different group. Statistics judge whether AGT can be as a early warning indicators of renal function decline.

ELIGIBILITY:
Inclusion Criteria:

* CKD, in the stage of 3 or 4, and kidney biopsy is preferred selection;
* Signed the informed consent;

Exclusion Criteria:

* Kidney cancer patients;
* Kidney transplantation;
* Hereditary kidney disease;
* Secondary renal disease(diabetic nephropathy and hypertensive nephropathy are excluded)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD（chronic kidney disease），in the stage of 3 or 4.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-02 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Urinary AGT level | 12 months
  Urinary AGT level can be an early bio-marker of intrarenal RAS activation and prewarning the deterioration of renal function.

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Department of Huashan Hospital, Shanghai, Shanghai Municipality, China